CLINICAL TRIAL: NCT00469820
Title: Posttransplant Immunotherapy With Donor Lymphocyte Infusions and Autologous Tumor Vaccines After HLA-Matched Transplant
Brief Title: Vaccine Therapy With or Without Donor Lymphocyte Infusion in Treating Patients With Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Multiple Myeloma Undergoing Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: J06118 CDR0000543531; P01CA015396 (NIH); P30CA006973 (NIH); JHOC-J06118
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Leukemia; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; stage III multiple myeloma; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; stage I multiple myeloma; stage II multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Congenital Abnormalities; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — FANG vaccine

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: peripheral blood lymphocyte therapy

SUMMARY:
RATIONALE: Vaccines made from the patient's cancer cells may help the body build an effective immune response to kill cancer cells. Giving vaccine therapy together with donor lymphocyte infusion after a stem cell transplant from the patient's brother or sister may kill any cancer cells that remain after transplant.

PURPOSE: This clinical trial is studying the side effects, best dose, and how well vaccine therapy with or without donor lymphocyte infusion works in treating patients with acute myeloid leukemia, acute lymphoblastic leukemia, or multiple myeloma undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine time to relapse and overall survival of patients with high-risk acute myeloid leukemia, acute lymphoblastic leukemia, or multiple myeloma treated with autologous tumor cell vaccine with or without donor lymphocyte infusion after HLA-matched related sibling nonmyeloablative hematopoietic stem cell transplantation.
* Evaluate the safety and tolerability of this regimen in these patients.
* Determine the maximum tolerated dose of donor lymphocyte infusions in these patients.

OUTLINE: Patients undergo collection of tumor cells for production of the cancer cell vaccine and then undergo HLA-matched related sibling nonmyeloablative hematopoietic stem cell transplantation (HSCT). Patients then receive cancer cell vaccine with or without donor lymphocyte infusion. The donor lymphocytes are obtained from the same relative who donated stem cells for the HSCT.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML), meeting any of the following criteria:

    * Relapsed disease
    * AML arising from myelodysplastic syndromes
    * Primary refractory disease
    * De novo AML with high-risk features
  * Acute lymphoblastic leukemia (ALL), meeting any of the following criteria:

    * De novo ALL that is Philadelphia chromosome positive or with t(4,11) cytogenetic features
    * Relapsed disease
  * Multiple myeloma (in need of treatment)
* Planning to undergo HLA-matched related sibling nonmyeloablative hematopoietic stem cell transplantation

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time to relapse
Overall survival
Safety and tolerability, in terms of incidence of graft-versus-host disease and local/systemic toxicities
Maximum tolerated dose of donor lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Huff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States